CLINICAL TRIAL: NCT02923180
Title: A Phase II Trial of Neoadjuvant Enoblituzumab (MGA271) in Men With Localized Intermediate- and High-Risk Prostate Cancer
Brief Title: Neoadjuvant Enoblituzumab (MGA271) in Men With Localized Intermediate and High-Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1693; IRB00103776 (Other: JHM IRB)
Record Dates: First submitted 2016-09-09; First posted 2016-10-04 (Estimated); Results first posted 2021-08-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: enobilituzumab
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enoblituzumab (Experimental): Men with localized intermediate and high-risk prostate cancer will be given neoadjuvant Enoblituzumab 15mg/kg IV weekly for 6 weeks followed by radical prostatectomy on day 50, with follow-up visits 30 days and 90 days post-prostatectomy. PSA values will be tracked for 3 years post-prostatectomy.
  Interventions: Drug: Enoblituzumab

INTERVENTIONS:
Drug: Enoblituzumab — Enoblituzumab 15mg/kg IV (in the vein) weekly for 6 doses beginning 50 days prior to radical prostatectomy.
  Other Names: MGA271

SUMMARY:
This study evaluates the safety, anti-tumor effect, and immunogenicity of Enoblituzumab given before radical prostatectomy. All patients will receive Enoblituzumab for 6 weekly doses beginning 50 days prior to radical prostatectomy.

DETAILED DESCRIPTION:
This is a single-center, single arm, open-label phase II study evaluating the safety, anti-tumor effect, and immunogenicity of neoadjuvant MGA271 given prior to radical prostatectomy in men with intermediate and high-risk localized prostate cancer. Eligible patients will receive MGA271 at a dose of 15mg/kg IV given weekly for 6 doses beginning 50 days prior to radical prostatectomy. 14 days after the last dose of MGA271, prostate glands will be harvested at the time of radical prostatectomy, and prostate tissue will be examined for the secondary endpoints. Follow-up evaluation for adverse events will occur 30 days and 90 days after surgery. Patients will then be followed by their urologists according to standard institutional practices, but will require PSA evaluations every 3 (±1) months during year 1 and every 6 (±2) months during years 2-3.

In Amendment 1, the study was expanded to enroll an additional 16 patients for a total of 32 patients to continue evaluating safety and better estimate the clinical benefit of Enoblituzumab in terms of undetectable PSA level (<0.1 ng/mL) at 12 months following radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate (clinical stage T1c-T3b, N0, M0) without involvement of lymph nodes, bone, or visceral organs
* Initial prostate biopsy is available for central pathologic review, and is confirmed to show at least 2 positive cores and a Gleason sum of ≥7
* Radical prostatectomy has been scheduled at Johns Hopkins Hospital
* Age ≥18 years
* ECOG performance status 0-1, or Karnofsky score ≥ 70% (see Appendix A)
* Adequate bone marrow, hepatic, and renal function:

  * WBC >3,000 cells/mm3
  * ANC >1,500 cells/mm3
  * Hemoglobin >9.0 g/dL
  * Platelet count >100,000 cells/mm3
  * Serum creatinine <1.5 × upper limit of normal (ULN)
  * Serum bilirubin <1.5 × ULN
  * ALT <3 × ULN
  * AST <3 × ULN
  * Alkaline phosphatase <3 × ULN
* The etiology of abnormal bilirubin and transaminase levels should be evaluated prior to study entry.
* Willingness to provide written informed consent and HIPAA authorization for the release of personal health information, and the ability to comply with the study requirements (note: HIPAA authorization will be included in the informed consent)
* Willingness to use barrier contraception from the time of first dose of MGA271 until the time of prostatectomy.

Exclusion Criteria:

* Presence of known lymph node involvement or distant metastases
* Other histologic types of prostate cancers such as ductal, sarcomatous, lymphoma, small cell, and neuroendocrine tumors
* Prior radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for prostate cancer
* Prior immunotherapy/vaccine therapy for prostate cancer
* Prior use of experimental agents for prostate cancer
* Concomitant treatment with other hormonal therapy or 5α-reductase inhibitors
* Current use of systemic corticosteroids or use of systemic corticosteroids within 4 weeks of enrollment (inhaled corticosteroids for asthma or COPD are permitted as are other non-systemic steroids such as topical corticosteroids)
* History or presence of autoimmune disease requiring systemic immunosuppression (including but not limited to: inflammatory bowel disease, systemic lupus erythematosus, vasculitis, rheumatoid arthritis, scleroderma, multiple sclerosis, hemolytic anemia, Sjögren syndrome, and sarcoidosis)
* History of malignancy within the last 3 years, with the exception of non-melanoma skin cancers and superficial bladder cancer
* Uncontrolled major active infectious, cardiovascular, pulmonary, hematologic, or psychiatric illnesses that would make the patient a poor study candidate
* Known prior or current history of HIV and/or hepatitis B/C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Shenderov, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shenderov E, De Marzo AM, Lotan TL, Wang H, Chan S, Lim SJ, Ji H, Allaf ME, Chapman C, Moore PA, Chen F, Sorg K, White AM, Church SE, Hudson B, Fields PA, Hu S, Denmeade SR, Pienta KJ, Pavlovich CP, Ross AE, Drake CG, Pardoll DM, Antonarakis ES. Neoadjuvant enoblituzumab in localized prostate cancer: a single-arm, phase 2 trial. Nat Med. 2023 Apr;29(4):888-897. doi: 10.1038/s41591-023-02284-w. Epub 2023 Apr 3. PMID 37012549

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 subjects signed consent to be screened for eligibility.
  - 1 subject signed consent, but did not meet the eligibility criteria to start the study (screen failure)
Period: Overall Study
Arm/Group | Enoblituzumab
Started | 32
Completed | 6
Not Completed | 26
Not completed — Off Study Due to Detectable PSA | 13
Not completed — Remaining in Long Term Follow Up for PSA | 13

BASELINE CHARACTERISTICS:
Population: Participants who met eligibility criteria
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Smoking History [Count of Participants; unit: Participants]
  Yes | 9
  No | 23
Family History of Prostate Cancer [Count of Participants; unit: Participants]
  Yes | 7
  No | 25
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased
  Participants
    0 | 31
    1 | 1
Body-mass index (kg/m^2) [Count of Participants; unit: Participants]
  Normal (BMI 18.5 - 24.9) | 6
  Overweight (BMI 25.0 - 29.9) | 14
  Obese (BMI ≥ 30.0) | 12
Gleason Group / Gleason sum at biopsy [Count of Participants; unit: Participants] — Gleason grade groups are defined as grade group 1 (Gleason score ≤ 6), grade group 2 (Gleason score 3+4=7), grade group 3 (Gleason score 4+3=7), grade group 4 (Gleason score 8), and grade group 5 (Gleason scores 9-10). A higher grade group reflects a worse outcome.
  Participants
    Grade Group 3: 4+3 | 5
    Grade Group 4: 4+4 | 8
    Grade Group 5: 4+5, 5+4, or 5+5 | 19
Previous Therapy [Count of Participants; unit: Participants] — Number of subjects who received therapy for prostate cancer prior to enrollment.
  Participants | 0
Stage T3 at initial diagnosis [Count of Participants; unit: Participants] — Stage T3 is defined as cancer growth outside of the prostate and possibly spread to the seminal vesicles.
  Participants
    Yes | 23
    No | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v4.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants
  Grade 1 | 31
  Grade 2 | 12
  Grade 3 | 4
  Grade 4 | 0

2. Primary Outcome: Efficacy of Neoadjuvant Enoblituzumab as Assessed by PSA0 Response Rate
Description: Number of participants with undetectable Prostate Specific Antigen (PSA <0.1 ng/mL) at 12 months following radical prostatectomy
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants
  PSA < 0.1 ng/mL | 21
  PSA ≥ 0.1 ng/mL | 11

3. Secondary Outcome: Quantify Markers of Apoptosis in Prostate Tumor Specimens of Treated Patients
Description: Quantify markers of apoptosis in prostate tumor specimens of treated patients using TUNEL staining and expressed as the mean staining percentage in tumor tissue
Time Frame: up to 5 years post-prostatectomy
Reporting Status: Not Posted

4. Secondary Outcome: Mean Staining Percentage of Markers of Cell Proliferation
Description: Quantify markers of cell proliferation in prostate tumor specimens of treated patients using Ki-67 staining and expressed by the mean staining percentage in tumor tissue
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable tissue samples.
Measure: Mean (Standard Deviation); unit: staining percentage
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
staining percentage | 11.92 (0.82)

5. Secondary Outcome: CD8+ T Cell Infiltration
Description: Mean staining percentage of CD8+ T-cells in harvested prostate glands from treated patients
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable tissue samples.
Measure: Mean (Standard Deviation); unit: staining percentage
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
staining percentage | 11.68 (0.71)

6. Secondary Outcome: PD-L1 Expression
Description: Mean staining percentage of PD-L1 in tumor tissue, assessed by immunohistochemistry (IHC) in the primary core specimens (pre-treatment) and the prostatectomy surgical specimens (post-treatment).
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable tissue samples.
Measure: Mean (Standard Deviation); unit: staining percentage
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
staining percentage | 10.66 (0.82)

7. Secondary Outcome: Regulatory T Cell (Treg) Infiltration
Description: Mean staining percentage of Treg cells in tumor tissue of treated patients, assessed through immunohistochemistry.
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable tissue samples.
Measure: Mean (Standard Deviation); unit: staining percentage
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
staining percentage | 9.36 (0.9)

8. Secondary Outcome: CD4+ T Cell Infiltration
Description: Mean staining percentage of CD4+ T-cells in tumor tissue of treated patients, assessed through immunohistochemistry.
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable tissue samples.
Measure: Mean (Standard Deviation); unit: staining percentage
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
staining percentage | 11.68 (0.71)

9. Secondary Outcome: Natural Killer (NK) Cell Density
Description: Mean staining percentage of NK cells in harvested prostate glands.
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable tissue samples.
Measure: Mean (Standard Deviation); unit: staining percentage
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
staining percentage | 11.92 (0.82)

10. Secondary Outcome: Enoblituzumab (MGA271) Drug Distribution Evaluated by Detection of MGA271 in Tumor Tissue
Description: Number of participants with positive or negative MGA271 detection in post-treatment prostate tumor specimens, as evaluated by IHC of fresh frozen sections.
Time Frame: 3 years
Population: The Overall Number of Participants Analyzed represents those evaluable for this outcome. Of the 32 participants who received study treatment, data from 2 subjects was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
Participants
  Positive | 28
  Negative | 2

11. Secondary Outcome: Pathological Complete Responses (pCR)
Description: Number of participants who achieve pCR, defined as absence of tumor identification on standard histological analysis of resected prostate specimens.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants | 0

12. Secondary Outcome: PSA Response Rates
Description: Number of participants with undetectable PSA (<0.1 ng/mL) at 3 months after prostatectomy.
Time Frame: 3 months post-prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants
  PSA <0.1 ng/mL | 26
  PSA ≥0.1 ng/mL | 6

13. Secondary Outcome: Time to PSA Recurrence
Description: Median time (months) from prostatectomy to time when PSA is ≥ 0.2 ng/mL. Estimated using Kaplan-Meier method.
Time Frame: up to 37 months post-prostatectomy
Measure: Median (Full Range); unit: months
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
months | 30 [3 to 37]

14. Secondary Outcome: Gleason Grade Group Change
Description: Number of participants with change in Gleason grade group from pre-treatment biopsy vs. post-treatment biopsy. "Downgrade" refers to a net grade group change less than zero, "upgrade" refers to net grade group change more than zero, and "no change" refers to stable Gleason grade group. Gleason grade groups are defined as grade group 1 (Gleason score ≤ 6), grade group 2 (Gleason score 3+4=7), grade group 3 (Gleason score 4+3=7), grade group 4 (Gleason score 8), and grade group 5 (Gleason scores 9-10).The lower the grade group, the better the outcome.
Time Frame: Day 50
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants
  Downgrade (< 0 net grade group change) | 16
  No Change (= 0 net grade group change) | 12
  Upgrade (> 0 net grade group change) | 4

15. Secondary Outcome: Number of Participants With PSA Percentage Decrease Prior to Radical Prostatectomy.
Description: The PSA percentage change is calculated as the difference from the PSA at day 50 prior to prostatectomy and PSA at screening. A negative value of PSA percentage change ("PSA percentage < 0") indicates a decrease in PSA from screening, and a positive value (PSA percentage change >= 0) indicates an increase in PSA from screening.
Time Frame: 50 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants
  PSA percentage change < 0 | 16
  PSA percentage change >= 0 | 16

16. Other Pre Specified Outcome: Androgen Receptor (AR) Quantification
Description: Mean staining percentage of AR in harvested prostate tissue, assessed by immunohistochemistry (IHC) staining for AR protein.
Time Frame: up to 3 years post-prostatectomy
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Tissue Androgen Concentrations
Description: Concentration (picogram/3 mg) of testosterone and 5α-dihydrotestosterone (DHT) in prostate tissue.
Time Frame: up to 3 years post prostatectomy
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Global Expression Profiling of Tumor Tissues
Description: Number of participants with changes in cellular composition, upregulation and downregulation of immune checkpoints, and other markers of activity versus exhaustion.
Time Frame: up to 3 years post-prostatectomy
Reporting Status: Not Posted

19. Other Pre Specified Outcome: IHC Analyses of CD137, CD16 and/or CD107A
Description: CD137, CD107A, and CD16 expression in prostate tumor specimens will be assessed by immunohistochemistry (IHC) in the prostatectomy surgical specimens (post-treatment). This endpoint will be expressed as the mean staining percentage of each of these in tumor tissue
Time Frame: up to 3 years post-prostatectomy
Reporting Status: Not Posted

20. Other Pre Specified Outcome: TCR Repertoire
Description: Fraction of peripherally expanded clones that are tumor associated for each participant.
Time Frame: 3 years post-prostatectomy
Population: Only 30 of the 32 participants enrolled in the trial had evaluable samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 30
Participants
  Number of participants with 100% peripheral expanded clones associated with tumor | 7
  Number of participants with 99% or less peripheral expanded clones associated with tumor | 23

21. Other Pre Specified Outcome: FC Receptor Genotyping
Description: Number of participants with CD16A, CD32A, and CD32B on Fc receptor.
Time Frame: up to 3 years post-prostatectomy
Reporting Status: Not Posted

22. Other Pre Specified Outcome: PBLs
Description: Number of participants with upregulation and downregulation of immune checkpoints and other markers of activity versus exhaustion, as assessed by flow cytometry at treatment day 1 (pre-treatment), treatment day 36 (post-treatment), and 30 days post-prostatectomy.
Time Frame: 3 years post-prostatectomy
Reporting Status: Not Posted

23. Other Pre Specified Outcome: B7-H3 Expression
Description: Number of participants with B7-H3 expression in prostate tumor specimens will be assessed by IHC (immunohistochemistry) in the primary core specimens (pre-treatment) and in the prostatectomy surgical specimens (post-treatment).
Time Frame: 3 years post-prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants | 28

24. Other Pre Specified Outcome: PD-1, LAG3, and TIM3 Expression
Description: PD-1, LAG3, and TIM3 expression in prostate tumor specimens will be assessed by IHC (immunohistochemistry) in the primary core specimens (pre-treatment) and in the prostatectomy surgical specimens (post-treatment). This endpoint will be expressed as the mean staining percentage in tumor tissue.
Time Frame: 3 Years post-prostatectomy
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Quantify Antigen-spread
Description: Number of participants with antigen-spread to on-target and off-target antigens.
Time Frame: 3 years post-prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 32
Participants
  Number of participants with IgG reactivity | 1
  Number of participants with IgM reactivity | 1
  Number of participants without antigen reactivity | 30

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Enoblituzumab
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enoblituzumab (N=32)
Infusion related reaction (Immune system disorders) | 1
Ascites (Blood and lymphatic system disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Cardiac Disorders - Other, Non-ST-Elevation, Myocardial Infarction (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoblituzumab (N=32)
Fatigue (General disorders) | 23 (34)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 5 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 31 (31)
Flu like symptoms (General disorders) | 13 (17)
Headache (Nervous system disorders) | 13 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9)
Edema limbs (General disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
White blood cell decreased (Investigations) | 1 (1)
Erectile dysfunction (Renal and urinary disorders) | 12 (12)
Creatinine increased (Investigations) | 3 (7)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Chills (General disorders) | 9 (10)
Vomiting (Gastrointestinal disorders) | 5 (5)
Fever (General disorders) | 8 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Serum amylase increased (Investigations) | 4 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Left knee weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipase increased (Investigations) | 2 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (10)
Infusion related reaction (General disorders) | 6 (7)
IV infiltration (Skin and subcutaneous tissue disorders) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Weight gain (Investigations) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Right eye stye (Eye disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Leukocyturia (Renal and urinary disorders) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Hematuria (Renal and urinary disorders) | 2 (2)
Lymphocele (Vascular disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Discolored urine (Renal and urinary disorders) | 1 (1)
Eye pain (Eye disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (2)
Myocarditis (Cardiac disorders) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (2)
Loss of dental filling (Surgical and medical procedures) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Left meniscus tear/injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Tachycardia (Vascular disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Incision site tenderness and erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT02923180/Prot_SAP_000.pdf